CLINICAL TRIAL: NCT04255901
Title: Efficacy of Head-point Acupuncture on Insomnia: A Prospective Case Series Study
Brief Title: Efficacy of Head-point Acupuncture on Insomnia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201900516A3
Record Dates: First submitted 2020-01-05; First posted 2020-02-05 (Actual); Last update posted 2020-07-14 (Actual); Status verified 2020-01

CONDITIONS: Sleep Initiation and Maintenance Disorders
Keywords: acupuncture; primary insomnia
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The investigators will conduct a single-center case series study. A total of 40 participants with insomnia will be enrolled. The aim of the study is to assess the therapeutic effect of head-point acupuncture for the treatment of insomnia.

DETAILED DESCRIPTION:
The investigators will conduct a single-center case series study. A total of 40 participants with insomnia will be enrolled, and will undergo GV20, EX-HN-1, GV21, GV22, GV23, GV24, GV29, and bilateral GB13 acupuncture treatment for 4 weeks.

The primary outcomes of therapeutic effect on insomnia are changes of the Pittsburgh Sleep Quality Index (PSQI), Epworth Sleepiness Scale (ESS), and the Hospital Anxiety and Depression Scale (HADS).The time frame of the three primary outcomes are: baseline week 0, week 2, week 4 and week 6.

The secondary outcomes of therapeutic effect on insomnia are sleep parameters including sleep efficiency (SE), sleep awakenings (SA) and total sleep time (TST) recorded by the actigraphy (time frame: baseline week 0, week 2, week 4 and week 6), as well as the heart rate viability(HRV) recorded by the ECG monitor (time frame: baseline week 0, week1, week 2, week 3, week 4 and week 6; and 30 minutes before and 60 minutes after acupuncture through study completion).

ELIGIBILITY:
Inclusion Criteria:

1. aged 20~80 years,
2. met the diagnostic criteria of insomnia according to the Diagnostic and Statistical Manual of Mental Disorders (Fifth Edition, DSM-V)
3. experienced insomnia at least three times a week for more than a month
4. voluntarily agreed with the investigation and signed a written informed con- sent form before the clinical trial started.

Exclusion Criteria:

1. a pregnant or lactating woman
2. the patient's insomnia is caused by mental disorders other than mild anxiety,
3. the patient has serious cardiovascular, liver, kidney or hematopoietic system disease
4. the patient's insomnia is caused by nervous system disease (eg, stroke, Parkinson's Disease)
5. the patient has taken Chinese herbs and herbal formulas for insomnia two weeks before the trial
6. the patient with cardiac pacemaker
7. the patient does not want to wear portable physiological signal recording device (SOMNOwatchTM) and handheld ECG monitor
8. the patient has a history of sleep apnea

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. aged 20~80 years,
  2. persistent difficulty in either falling asleep, remaining asleep through the night, or waking up too early at least three nights a week for more than a month, and not suffered from any secondary diseases.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2020-08-01 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Changes of The Epworth sleepiness scale (ESS) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The Epworth sleepiness scale (ESS) containing eight items that ask for self-reported disclosure of the expectation of "dozing" in a variety of situations. A sum of responses is calculated for a total score ranging from 0 to 24, higher scores mean a worse outcome.
Changes of The HADS(The Hospital Anxiety and Depression Scale) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The Hospital Anxiety and Depression Scale is a 14-items self-administered questionnaire, the scores ranged from 0 to 21 for anxiety and 0 to 21 for depression, higher scores mean a worse outcome.
Changes of The PSQI(Pittsburgh Sleep Quality Index) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The 19 questions are combined into seven clinically-derived component scores, each weighted equally from 0-3. The seven component scores are added to obtain a global score ranging from 0-21, with higher scores indicating worse sleep quality.

SECONDARY OUTCOMES:
HRV(Heart rate viability) | Baseline week 0, week1, week 2, week 3, week 4 and week 6; and 30 minutes before and 60 minutes after acupuncture through study completion, an average of 1 year.
  Frequency-domain analysis of heart rate variability (HRV), a noninvasive method, has been used to reflect cardiac autonomic nervous activity in humans. The high-frequency power (HF; 0.15-0.4 Hz) of HRV represents vagal (parasympathetic) control of heart rate. The low-frequency power (LF; 0.04- 0.15 Hz) of HRV is jointly contributed by both sympathetic and vagal nerves, whereas normalized LF (nLF) is regarded as the sympathetic modulation.
actigraphy (3-day) | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  Actigraphy provides objective estimates of sleep parameters including: SE(sleep efficiency), SA(sleep awakenings), TST(total sleep time)
sleep diary | Baseline week 0, week 2, week 4 & 2 weeks post-tx (week 6)
  The sleep diary provides daily subjective estimates of sleep parameters including: daytime nap, sleep aids intake, bedtime, sleep onset latency, frequency of nocturnal awakenings, awakenings duration, wake-up time, arising time, feeling upon arising (five-point scale) and sleep quality (five-point scale).

IPD SHARING:
Plan to Share IPD: No
There will be a research number representing the identity. This number will not display the name, identification number, and address.
  For the results and diagnosis of the visit, the research host will maintain a confidential attitude and carefully maintain the privacy. If research results are published, the identity will remain confidential.
  Please also understand that if the participant signs the consent form, the participant agrees that the visit record can be directly reviewed by the monitor, auditor, research ethics committee and the competent authority to ensure that the research process and data comply with relevant laws and regulations. These people also promise not to violate the confidentiality of your identity.